CLINICAL TRIAL: NCT02637518
Title: A Comprehensive Validation of Frailty Assessment Tools to Screen and Diagnose Frailty in Different Clinical and Social Settings and to Provide Instruments for Integrated Care in Older Adults.
Brief Title: Comprehensive Validation of Frailty Assessment Tools in Older Adults in Different Clinical and Social Settings
Acronym: FRAILTOOLS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Getafe (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: 662887
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Syndrome
Keywords: Frailty; Frailty screening tools; Clinical settings; Social settings; Geriatrics; Functional autonomy; Disability
MeSH Terms: conditions — Syndrome; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Hospital Universitario de Getafe: Assessment of frailty tools in elderly people
  The Geriatric Department attends patients:
  1800/year - acute unit. 800/year - Orthogeriatrics and Interconsultation Unit. 300/year - Day Hospital. 4000/year - Outpatient office. 1200/year - Domiciliary Care.
  Interventions: Other: Assessment of frailty tools in elderly people
- Diabetes Frail Ltd.: Assessment of frailty tools in elderly people Has significant experience in managing research studies in older people.
  Interventions: Other: Assessment of frailty tools in elderly people
- Università Cattólica del Sacro Cuore: Assessment of frailty tools in elderly people
  The Geriatric Unit is compounded by:
  24 beds of Acute Care Ward 46 beds of Intensive Rehabilitation Unit 20 beds of Day Hospital Outpatient clinic
  Interventions: Other: Assessment of frailty tools in elderly people
- Gérontopole de Toulouse: Assessment of frailty tools in elderly people
  The Geriatric Unit is compounded by:
  5 Acute Care Units - 100 beds. 3 Rehabilitation Unit - 75 beds. Long term care Unit - 140 beds. 2 Day Hospitals Outpatient Clinic
  Interventions: Other: Assessment of frailty tools in elderly people
- Jagiellonian University Medical College: Assessment of frailty tools in elderly people The Department of Internal Medicine and Gerontology is the largest centre in Poland limited to the Geriatric market.
  Interventions: Other: Assessment of frailty tools in elderly people

INTERVENTIONS:
Other: Assessment of frailty tools in elderly people — Assessment of the tools as screening/diagnosis instruments in older adults attended in Primary Care. To build the integration of tools in algorithms to be used in each setting of care and along the settings to permit an integrated care in different conditions (isolated assessment or sequential assessment)

SUMMARY:
There is a proved strong evidence of the usefulness of frailty as a predictive factor of relevant and desired outcomes in populations of older adults. Several studies have been published showing the utility of the concept in improving the prognosis accuracy and the prediction of different risks (hospitalisations, surgical and non surgical complications, length of stay, death, incident disability, etc.) in emergency departments, surgical patients, and inpatients with cardiovascular disease. The studies have placed the focus in assessing population risk, while the validation process for these instruments as diagnosis or screening tools has been usually neglected. FRAILTOOLS aims to assess the usefulness as screening and diagnosis tools of some selected instruments to detect frailty in both clinical (Hospital and Primary Care) and social (Nursing Homes) settings, providing diagnostic algorithms clinically sound. Target groups are all of those older adults at risk of frailty (pre-frail) plus those that are frail and are at risk for developing disability. According to the published prevalence of these two conditions, the target population concerned by this project represents around 40-50% of people older than 65, and 60-70% of people older than 75. Once determining the best tools of screening and diagnosis in different settings of care, investigators will research conclusions of these people wherever the level of care they need and currently use. The benefit will spend to the Health System and Social Care as it will provide validated instruments that are necessary to provide an appropriate care for older adults by means of a comprehensive, continued, coordinated and integrated care.

DETAILED DESCRIPTION:
Quality assurance plan:

According to the European's Commission guidelines, the procedure for quality control focuses on the deliverables revision and in the quality of each procedure. The deliverables will be sent to the Administrative committee. The administrative Committee, composed by the Project's Promoter and its associates, will assume the role as a quality manager. It includes the following tasks:

Making sure of the monitoring of all of the changes in documentation. Making sure the activity's coordination and reports are completed according to an adequate quality and in an appropriate manner.

Reviewing the contract deliverables. Monitoring and auditing the project's activities according to plan, making the specific revisions of the contractual deliverables, directed to the achievement of the established objectives.

The electronic Case Report Form (eCRF) has been designed to capture all data required in the protocol. A unique eCRF will be completed for subject, taking into account the protection law in each country of the study.Subjects will be identified by a unique subject number (with key held by the relevant partner), so none identification card number will be recorded on the eCRF or the database. The monitor will guarantee that the eCRF is fully and correctly fill up according to the source documents. The researcher will assure that all data recorded in the eCRF coincide with the information recorded in the source documents.

Plan for missing data to address situations where variables are reported as missing:

The investigators will check the missing data in each eCRF and source documents.

Statistical analysis:

Investigator will assess the associations of each scale with the outcome for each setting and outcome through logistic regressions. First, investigators will compute the classification performance (sensitivity, specificity, Receptors Operational Curve (ROC), Area Under the Curve (AUC), predictive values, likelihood ratios) for each model. Second, investigators will study the feasibility of the models taking into account the time needed for the scale and the percentage of patients that can be assessed per case. Investigators will evaluate the sensitivity to change of the scales and the covariance of the scales with other measures as the SPPB through a mixed linear model.

Sample Size: Participants will be recruited in Spain, Italy, France, United Kingdom and Poland. The total sample will be of 1.940 subjects. Each participating centre will have to recruit a total of 388 patients, corresponding to 97 subjects in each clinical setting by centre.

ELIGIBILITY:
Inclusion Criteria:

* People older than 75 years old, who sign the informed consent after accepting their participation.

Exclusion Criteria:

* General exclusion criteria will be an MMSE score less than 20 points or having a terminal illness (life expectancy < 6 months).
* Subjects included from the hospital ward (Acute Geriatric Unit and Outpatient
* Geriatric Consultation) and primary care will have additional exclusion criteria: dependency in more than 2 Instrumental Activities of Daily Living (IADL) in women (Lawton < 6), and in more than 3 IADL in men (Lawton < 5).
* Subjects seen in a nursing home setting will be excluded if they obtain less than 40 points in the Barthel index.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: People older than 75 years old will be included, recruited from different clinical settings such as clinical (hospital or primary care) and social (nursing homes).
Sampling Method: Non-Probability Sample
Enrollment: 1940 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-08 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Mortality | 18 months
  data obtained from the official registration of the country of the corresponding partner. When not available, other methods will be used (asking to a proxy, calls to nursing homes, medical registries, etc.).
Functional disability | 18 months
  Defined as a loss of at least one point in the Short Physical Performance Battery (SPPB).
Disability to perform IADL | 18 months
  Defined as a loss of at least one point in the Lawton Index
Disability to perform BADL | 18 months
  Defined as a loss of at least one point in the Barthel Index.
Falls | 18 months
  Data will be collected by the participant's verbal recall (self-assessed) and will be registered in the electronic Case Report Form (eCRF).
Incident cognitive impairment | 18 months
  Defined by a reduction of 2 or more points in the Mini-Mental State Examination (MMSE).

SECONDARY OUTCOMES:
Frailty classification performance | 18 months
  Performance of the instruments by clinical setting: six frailty assessment tools will be used in four different levels of care. The performance of each scale in the classification of frailty will be established.
Tool feasibility | 18 months
  Composed by two main conditions: the percentage of people that are assessed by each tool in each setting (adequacy) and the time for carrying out the the tool assessment.
Sensitivity to change in frailty status | 18 months
  Evaluate the changes in the assessment level of patients observed at 12 and 18 months with each of the tools and their correlations with the changes observed in the patient´s functional status.
Qualification as a screening and/or diagnosis tool | 18 months
  Evaluate the utility of each scale as a frailty detection method for screening or diagnosis, using pre-established criteria.

CONTACTS AND LOCATIONS:
Overall Officials: LEOCADIO RODRIGUEZ MAÑAS, MD, PhD, Principal Investigator — HOSPITAL UNIVERSITARIO DE GETAFE
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Rodriguez-Manas L, Fried LP. Frailty in the clinical scenario. Lancet. 2015 Feb 14;385(9968):e7-e9. doi: 10.1016/S0140-6736(14)61595-6. Epub 2014 Nov 6. No abstract available. PMID 25468154
- [Background] Rodriguez-Manas L, Sinclair AJ. Frailty: the quest for new domains, clinical definitions and subtypes. Is this justified on new evidence emerging? J Nutr Health Aging. 2014 Jan;18(1):92-4. doi: 10.1007/s12603-013-0433-9. No abstract available. PMID 24402396
- [Background] Garcia-Garcia FJ, Carcaillon L, Fernandez-Tresguerres J, Alfaro A, Larrion JL, Castillo C, Rodriguez-Manas L. A new operational definition of frailty: the Frailty Trait Scale. J Am Med Dir Assoc. 2014 May;15(5):371.e7-371.e13. doi: 10.1016/j.jamda.2014.01.004. Epub 2014 Mar 2. PMID 24598478
- [Background] Gill TM, Gahbauer EA, Allore HG, Han L. Transitions between frailty states among community-living older persons. Arch Intern Med. 2006 Feb 27;166(4):418-23. doi: 10.1001/archinte.166.4.418. PMID 16505261
- [Background] Fried LP, Guralnik JM. Disability in older adults: evidence regarding significance, etiology, and risk. J Am Geriatr Soc. 1997 Jan;45(1):92-100. doi: 10.1111/j.1532-5415.1997.tb00986.x. PMID 8994496
- [Derived] Oviedo-Briones M, Rodriguez-Laso A, Carnicero JA, Gryglewska B, Sinclair AJ, Landi F, Vellas B, Rodriguez Artalejo F, Checa-Lopez M, Rodriguez-Manas L. The ability of eight frailty instruments to identify adverse outcomes across different settings: the FRAILTOOLS project. J Cachexia Sarcopenia Muscle. 2022 Jun;13(3):1487-1501. doi: 10.1002/jcsm.12990. Epub 2022 Apr 15. PMID 35429109
- [Derived] Checa-Lopez M, Oviedo-Briones M, Pardo-Gomez A, Gonzales-Turin J, Guevara-Guevara T, Carnicero JA, Alamo-Ascencio S, Landi F, Cesari M, Grodzicki T, Rodriguez-Manas L; FRAILTOOLS consortium. FRAILTOOLS study protocol: a comprehensive validation of frailty assessment tools to screen and diagnose frailty in different clinical and social settings and to provide instruments for integrated care in older adults. BMC Geriatr. 2019 Mar 18;19(1):86. doi: 10.1186/s12877-019-1042-1. PMID 30885132